CLINICAL TRIAL: NCT00568035
Title: Phase II Study of QR-333 for the Treatment of Symptomatic Diabetic Peripheral Neuropathy
Brief Title: Safety and Efficacy Study of QR-333 in Patient's With Symptomatic Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Quigley Pharma, Inc. (Industry)
Responsible Party: Quigley Pharma, Inc., Richard Rosenbloom
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QR-333-002
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Last update posted 2009-01-08 (Estimated); Status verified 2009-01

CONDITIONS: Diabetic Neuropathy
Keywords: diabetic; peripheral; neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- QR-333 (Active Comparator)
  Interventions: Drug: QR-333
- Placebo (Placebo Comparator)
  Interventions: Drug: QR-333

INTERVENTIONS:
Drug: QR-333 — QR-333 or placebo will be applied three times a day for 12 weeks

SUMMARY:
The purpose of this study is to determine whether QR-333 is safe and effective in the treatment of diabetic neuropathy as compared to placebo.

DETAILED DESCRIPTION:
Diabetic neuropathy is among the most common complication of diabetes, resulting in pain and numbness, which affects the patients sleep, functioning and well-being. The pain is often accompanied by unpleasant sensations described as buzzing, cramp-like, burning, or jolting. The pain is usually symmetrical and occurs in the upper and lower extremities following a "glove and stocking" distribution.

To date there is no fully effective treatment for diabetic neuropathy. Therapy is tailored individually according to subject complaints and may be selected from categories including Non-steroidal anti-inflammatory drugs (NSAIDs) and adjuvant analgesics (including tricyclic antidepressants and anticonvulsants).

The clinical trial is being conducted to determine the safety and efficacy of QR-333 in the treatment of diabetic neuropathy as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of diabetic neuropathy
* must have some pain daily in the lower limbs due to diabetic polyneuropathy for at least 3 months prior to enrollment
* must be willing to comply with study directions, write information in a diary (such as pain medications taken), read and comprehend written instructions, complete questionnaires, and have the ability to apply the cream as directed

Exclusion Criteria:

* uncontrolled pain that has persisted for > 12 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Determine the safety of a three times daily application of QR-333 as compared to placebo. | 12 Weeks

SECONDARY OUTCOMES:
Determine the efficacy of QR-333 on symptoms of diabetic neuropathy and the impact of QR-333 on the daily activities (including pain and sleep disturbance) of subjects with symptomatic diabetic neuropathy as compared to placebo. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philip Raskin, MD, Study Chair — University of Texas, Southwestern Medical Center at Dallas
Locations (19):
- United States (19):
  - Parkway Medical Center, Birmingham, Alabama
  - Seale Harris Clinic / Alliance Clinical Research, Birmingham, Alabama
  - Pacific Sleep Medicine Services, Inc, Fountain Valley, California
  - Advanced Medical Research, LLC, Lakewood, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Renstar Medical Research, Ocala, Florida
  - Baptist Clinical Research, Pensacola, Florida
  - Stedman Clinical Trails, Tampa, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - A&A Pain Institute, St Louis, Missouri
  - Rwjms/Umdnj, New Brunswick, New Jersey
  - Land Clinical Studies, West Caldwell, New Jersey
  - Kaleida Health, Diabetes Center of WNY, Buffalo, New York
  - ECU Diabetes Research Center, Brody School of Medicine, Greenville, North Carolina
  - Hartwell Research Group / Anderson Family Care, Anderson, South Carolina
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - dgd Research, San Antonio, Texas
  - Endeavor Clinical Trials, PA, San Antonio, Texas
  - Rainier Clinical Research Center, Inc, Renton, Washington